CLINICAL TRIAL: NCT00601458
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Pregabalin and Naproxen Sodium on Postoperative Pain After Bunionectomy
Brief Title: Bunionectomy Study (0000-063)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-063; 063; 2007_661
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Results first posted 2010-04-08 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-03

CONDITIONS: Acute Pain
Keywords: Primary, unilateral, first metatarsal bunionectomy with osteotomy
MeSH Terms: conditions — Acute Pain | interventions — Pregabalin; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Arm 1: Pregabalin 300 mg (Active Comparator)
  Interventions: Drug: pregabalin
- Arm 2: naproxen sodium 550 mg (Active Comparator)
  Interventions: Drug: naproxen sodium
- Arm 3: Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: pregabalin — Patients will be randomized just prior to surgery to 1 of 3 study treatments: pregabalin (300 mg) treatment will be administered approximately 1 hour prior to surgery. Postoperatively, pregabalin (150 mg) will be dosed starting at 8 hours following T=0 and every 8 hours until 40 hours following T=0.
  Arms: Arm 1: Pregabalin 300 mg
Drug: naproxen sodium — Patients will be randomized just prior to surgery to 1 of 3 study treatments: naproxen sodium (550 mg) treatment will be administered approximately 1 hour prior to surgery. Postoperatively, naproxen sodium will be dosed starting 12 hours following T=0 and every 12 hours until 36 hours following T=0.
  Other Names: naproxen
  Arms: Arm 2: naproxen sodium 550 mg
Drug: Comparator: Placebo — Patients will be randomized just prior to surgery to 1 of 3 study treatments: placebo treatment will be administered approximately 1 hour prior to surgery. Postoperatively, placebo will be dosed starting at 8 hours following T=0 and every 8 hours until 40 hours following T=0.
  Arms: Arm 3: Placebo

SUMMARY:
We are interested in whether bunionectomy can be used as a model to study the treatment of acute pain. It has been used to study the effect of Non-Steroidal Anti-inflammatory (NSAIDS) medications (such as ibuprofen) and other pain relieving drugs. We are interested to know if this model is useful to study other drugs for the treatment of acute pain. The other drugs being tested in this study are pregabalin and naproxen sodium. These drugs are approved for use by the Food and Drug Administration (FDA). This study is designed to test whether these two drugs are effective in treating pain after a bunionectomy.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a man or woman between 18 and 65 years of age
* For Women of Child-bearing potential: woman who is currently not pregnant not nursing and who is willing to use a medically acceptable method of birth control from the time after the screening visit until completion of the follow-up visit
* Patient is scheduled to have a bunionectomy
* Patient must be willing to stay at the study site throughout the 48-hour observation period following surgery and is willing to complete a 2-week follow up
* Patient is capable of operating a Patient Controlled Analgesia device

Exclusion Criteria:

* Patient is being treated for a disease and has not been on a stable dose of medication for at least 2 weeks prior to surgery
* Patient has used or intends to use any of the medications that are prohibited by the protocol, which could interfere with the evaluation of the study drugs
* Patient has an estimated creatinine clearance of < or = 60 mL per min
* Patient has a history of drug abuse or dependence, or patient has a positive urine drug screen
* Patient has a condition that prevents clear communication concerning pain perception (such as diabetic neuropathy, peripheral neuropathy, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Wang H, Gargano C, Lukac S, Jackson A, Beals C, Smiley P, Drexel M, Ruddy M, Herman G, Johnson-Levonas AO, Medve R, Webster L, Reicin A. An enhanced bunionectomy model as a potential tool for early decision-making in the development of new analgesics. Adv Ther. 2010 Dec;27(12):963-80. doi: 10.1007/s12325-010-0084-8. Epub 2010 Nov 3. PMID 21052881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 25 July 2007
  Last Patient Last Visit: 28 January 2008
  1 site
Groups:
- Pregabalin 300 mg: Active Comparator: Arm 1: Pregabalin 300 mg
  Pregabalin (300 mg) treatment was administered approximately 1 hour prior to surgery. Postoperatively, pregabalin (150 mg) was dosed starting at 8 hours following T=0 and every 8 hours until 40 hours following T=0.
- Naproxen Sodium 550 mg: Active Comparator: Arm 2: Naproxen sodium 550 mg
  Naproxen sodium (550 mg) treatment was administered approximately 1 hour prior to surgery. Postoperatively, naproxen sodium was dosed starting at 12 hours following T=0 and every 12 hours until 36 hours following T=0.
- Placebo: Placebo treatment was administered approximately 1 hour prior to surgery. Postoperatively, placebo was dosed starting at 8 hours following T=0 and every 8 hours until 40 hours following T=0.
Period: Overall Study
Arm/Group | Pregabalin 300 mg | Naproxen Sodium 550 mg | Placebo
Started | 36 | 34 | 30
Completed | 32 | 29 | 28
Not Completed | 4 | 5 | 2
Not completed — Dosing Error | 1 | 0 | 0
Not completed — Incomplete Data | 0 | 2 | 0
Not completed — Protocol Violation | 3 | 2 | 1
Not completed — Early Termination | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin 300 mg | Naproxen Sodium 550 mg | Placebo | Total
Number analyzed (Participants) | 32 | 29 | 28 | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (14.1) | 40.6 (13.5) | 38.8 (11.6) | 39.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 23 | 73
  Male | 5 | 6 | 5 | 16
Body Weight [Mean (Standard Deviation); unit: Kilograms] | 72.3 (18.1) | 76.7 (17.2) | 77.2 (16.9) | 75.3 (17.4)
Lidocaine Use [Mean (Standard Deviation); unit: Milliliters] — Regional anesthesia required during surgery
  Milliliters | 15.0 (2.3) | 15.9 (2.7) | 14.6 (1.6) | 15.2 (2.2)
Propofol Use [Mean (Standard Deviation); unit: Milligrams] | 348.4 (132.9) | 364.5 (122.8) | 353.9 (105.8) | 355.4 (121.1)

OUTCOME MEASURES:

1. Primary Outcome: Total Patient Controlled Analgesic (PCA) Hydromorphone Consumption Over the 24 Hours Post-surgery
Description: Total dose (amount) of hydromorphone via patient controlled analgesic (PCA) pump required in the 24 hours post-surgery in each of the treatment arms: placebo, pregabalin 300 mg or naproxen 550 mg.
Time Frame: First 24 hours following surgery
Measure: Geometric Mean (Inter-Quartile Range); unit: milligrams
Arm/Group | Pregabalin 300 mg | Naproxen Sodium 550 mg | Placebo
Number analyzed (Participants) | 32 | 29 | 28
milligrams | 2.94 [2.00 to 5.35] | 2.07 [0.80 to 4.60] | 5.96 [4.50 to 7.70]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA — 1-sided alpha = 0.045 Hochberg closed testing procedure; Mean Difference (Final Values) = -50.7, 97.8% CI [-73.6 to -8.0] — The natural log scale treatment difference (pregabalin - placebo) and 97.8% CI for the treatment difference were exponentiated and reported as a percentage reduction in 24-h cumulative hydromorphone consumption
Statistical Analysis 2: Comparison: Naproxen Sodium 550 mg vs Placebo; Test type: Superiority or Other; p = 0.0001, ANOVA — 1-sided alpha = 0.045 Hochberg closed testing procedure; Mean Difference (Final Values) = -65.4, 97.8% CI [-81.7 to -34.6] — The natural log scale treatment difference (naproxen - placebo) and 97.8% CI for the treatment difference were exponentiated and reported as a percentage reduction in 24-h cumulative hydromorphone consumption

2. Secondary Outcome: Time to First Request of PCA Hydromorphone
Description: Time (in hours) to first patient controlled analgesic (PCA) pump use after surgery in each of the treatment arms: placebo, pregabalin 300 mg or naproxen 550 mg.
Time Frame: First 24 hours following surgery
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Pregabalin 300 mg | Naproxen Sodium 550 mg | Placebo
Number analyzed (Participants) | 32 | 29 | 28
Hours | 7.3 [5.8 to 9.4] | 9.1 [7.1 to 13.6] | 5.8 [5.1 to 7.4]
Statistical Analysis 1: Comparison: Pregabalin 300 mg vs Placebo; Test type: Superiority or Other; p = 0.004, Log Rank — 1-sided alpha = 0.045 Hochberg closed testing procedure; Median Difference (Final Values) = 1.46, 95% CI [0.183 to 2.95] — Hodges-Lehmann procedure was used to obtain an estimate of the difference in medians and an exact CI for the difference in medians
Statistical Analysis 2: Comparison: Naproxen Sodium 550 mg vs Placebo; Test type: Superiority or Other; p < 0.001, Log Rank — 1-sided alpha = 0.045 Hochberg closed testing procedure; Median Difference (Final Values) = 3.70, 95% CI [1.77 to 6.72] — [estimate comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: AEs were collected from the time the subject signed consent until 14 days following the last dose of study mediciation.
Description: AE were assessed by clinical evaluation including vital signs, physical examination. medical history, clinical laboratory safety assessment (chemistry, hematology, urinalysis) and ECG at time points specified in the study. Subjects were queried at each visit for any clinical adverse experiences that may have occurred since the previous visit.
Arm/Group | Pregabalin 300 mg | Naproxen Sodium 550 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/34 | 0/30
Other Adverse Events (participants affected / at risk) | 26/36 | 19/34 | 25/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 300 mg (N=36) | Naproxen Sodium 550 mg (N=34) | Placebo (N=30)
Vision Blurred (Eye disorders) | 0 | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 16 | 14 | 21
Vomiting (Gastrointestinal disorders) | 7 | 9 | 18
Chills (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Blood Pressure Decreased (Investigations) | 1 | 0 | 0
Oxygen Saturation Decreased (Investigations) | 2 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 6 | 5 | 3
Headache (Nervous system disorders) | 8 | 1 | 4
Somnolence (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Vulvovaginal Dryness (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Blood Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 5 | 5
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.